CLINICAL TRIAL: NCT05386173
Title: Effect of Fetal Aortic Valvuloplasty on Outcomes. A Prospective Observational Cohort Study With a Comparison Cohort
Brief Title: Effect of Fetal Aortic Valvuloplasty on Outcomes
Acronym: FASSprosp
Status: Recruiting | Type: Observational
Sponsor: Queen Silvia Children's Hospital, Gothenburg, Sweden (Other)
Collaborators: Swedish Heart Lung Foundation (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Mellander, Associate professor, Consultant pediatric and fetal cardiology, Queen Silvia Children's Hospital, Gothenburg, Sweden
Other Study IDs: FASSprosp
Record Dates: First submitted 2022-05-13; First posted 2022-05-23 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Congenital Heart Disease; Aortic Valve Stenosis; Fetal Cardiac Disorder; Hypoplastic Left Heart Syndrome
MeSH Terms: conditions — Heart Defects, Congenital; Aortic Valve Stenosis; Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fetal intervention group: Fetuses with aortic valve stenosis satisfying all of the inclusion/exclusion criteria
  Interventions: Procedure: Fetal aortic balloon dilatation
- Fetal non-intervention group: Fetuses with aortic valve stenosis satisfying all of the inclusion/exclusion criteria which are identical with the criteria in the Fetal intervention group

INTERVENTIONS:
Procedure: Fetal aortic balloon dilatation — Fetal valvuloplasty will be performed as described in Arzt W, Wertaschnigg D, Veit I, Klement F, Gitter R, Tulzer G. Intrauterine aortic valvuloplasty in fetuses with critical aortic stenosis: experience and results of 24 procedures. Ultrasound Obstet Gynecol. 2011;37:689-695. with minor variations between centers involved. Technical success is defined as improved forward flow and/or new aortic regurgitation.
  Groups: Fetal intervention group

SUMMARY:
In one of the most severe congenital heart defects, hypoplastic left heart syndrome (HLHS), the left ventricle is underdeveloped and the prognosis is worse than in most other heart defects. The underdevelopment can occur gradually during fetal growth caused by a narrowing of the aortic valve. At some international centers, such fetuses are treated with a balloon dilation of the narrowed valve, but there is no scientifically sound evidence that this treatment is effective.

The aim of this study is: 1/ to evaluate whether balloon dilation during the fetal period of a narrowed aortic valve can reduce the risk of the left ventricle becoming underdeveloped and the baby being born with a so-called univentricular heart (HLHS); 2/ to investigate whether such treatment improves the prognosis for this group of children with a very complex and severe heart defect and 3/ to also describe side effects and risks in fetuses and mothers of the fetal procedure.

DETAILED DESCRIPTION:
Routinely collected pre- and postnatal clinical data will be entered into a digital database and echocardiographic examinations will be uploaded to a server. A core lab will measure and analyze all echocardiographic examinations according to protocol. The growth of the left heart structures and the postnatal outcome will be compared between the intervention and non-intervention groups.

The decision whether a fetal balloon dilatation shall be attempted is not part of the study protocol. The number of examinations of mother/fetus/infant in this study is not different from the number of examinations that will be recommended for someone choosing not to be part of this study. Participation in the study does not affect the care and treatment mothers and fetuses are receiving during pregnancy, nor how the infant is examined and treated after birth.

ELIGIBILITY:
Inclusion Criteria:

A. All of the following echocardiographic criteria need to be satisfied between 23+0 and 31+6 weeks (z-scores according to Schneider et al):

1. Aortic valve stenosis with antegrade flow through the valve
2. Predominantly left-to-right shunt at the atrial level
3. Predominantly retrograde flow in the aortic arch between the first two brachiocephalic vessels
4. Qualitatively depressed left ventricular function
5. Left ventricular end-diastolic diameter Z-score > ±0
6. Left ventricular inlet length in diastole :

   1. Gestational age ≤ 24+6: Z-score > ±0
   2. Gestational age 25+0 to 27+6: Z-score > -0.75
   3. Gestational age ≥ 28+0: Z-score > -1.50
7. Mitral valve diameter in diastole Z-score > -2.0

B. All of the following postnatal treatment options need to be available: 1. Surgical or catheter based aortic valvotomy 2. Ross-Konno surgery 3. Norwood or hybrid stage-one surgery

Exclusion Criteria:

1. Any associated cardiac defect except persistent left superior vena cava and coarctation of the aorta
2. Any significant (i.e. that might influence outcome) extracardiac anomaly and/or known chromosomal aberration. Also, if such a condition is present at inclusion but diagnosed only after birth the case will be retrospectively excluded.

Ages: 23 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of fetuses and children with aortic valve stenosis and/or hypoplastic left heart syndrome
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Transplantation-free survival | Follow-up from study inclusion during fetal life until 2 years postnatal age
  Transplantation-free survival from fetal diagnosis to 2 years postnatal age with a biventricular circulation without pulmonary hypertension at that time. Absence of pulmonary hypertension is defined as a TR max velocity ≤ 2.8 m/s with no other echocardiographic signs of pulmonary hypertension and/or catheter data showing a mean pulmonary arterial pressure <25 mmHg.

SECONDARY OUTCOMES:
Intervention-related fetal death | From the time of fetal intervention until 24 hours after the intervention
  Intervention-related fetal death (defined as fetal death within 24 hours of procedure)
Fetal death not directly related to the intervention | From 24 hours after fetal intervention until fetal death, up to 20 weeks after study inclusion.
  Fetal death not directly related to the intervention, except termination of pregnancy
Maternal complications to fetal intervention procedure | From time of fetal intervention until 24 hours after the intervention
  Maternal complications to procedure requiring intensive care or resulting in maternal death
Preterm delivery | From time of fetal intervention until 37 weeks gestational age, maximum 14 weeks
  Preterm delivery before 37 weeks gestational age
Fetal left heart growth | From the date of study inclusion until just before the first postnatal catheter or surgical intervention, or death, whichever comes first, total time frame 7 months
  Fetal left heart growth as measured with dimensions expressed a z-scores of the mitral valve diameter, left ventricular inlet length and aortic valve diameter

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - Fetal Cardiovascular Program, University of California San Francisco, San Francisco, California
  - Congenital Heart Collaborative, Nationwide Children's Hospital, Columbus, Ohio
- Kinderherzzentrum Linz, Linz, Austria
- The Hospital for Sick Children Toronto, Toronto, Canada
- Department of Paediatric Cardiology, Helsinki University Children's Hospital, Helsinki, Finland
- Germany (3):
  - Pediatric Cardiology - University Hospital Bonn, Bonn
  - Department of Pediatric and Congenital Cardiology, University of Heidelberg, Heidelberg
  - University hospital Technical university, mother- and-child center, Munich
- Department of Perinatal Cardiology and Congenital Anomalies, Centre of Postgraduate Medical Education., Warsaw, Poland
- Fetal Medicine Unit, Dept. Obstetrics & Gynecology University Hospital 12 de Octubre, Madrid, Spain
- Sweden (3):
  - Department of Pediatric Cardiology, Skane University Hospital, Lund
  - Department of pediatric cardiology, Karolinska Institute, Stockholm
  - Department of Pediatrics, Umeå University Hospital, Umeå

IPD SHARING:
Plan to Share IPD: No